CLINICAL TRIAL: NCT05258266
Title: A Dose-Escalation and Expansion Phase I/IIa Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of ZX-101A Monotherapy in Patients With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Activity, Safety and Tolerability of ZX-101A in Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing Zenshine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZX-101A-201
Record Dates: First submitted 2022-01-27; First posted 2022-02-28 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- ZX-101A Dose Level A (Experimental): ZX-101A administered orally at level A once daily in a 28-day cycle
  Interventions: Drug: ZX-101A
- ZX-101A Dose Level B (Experimental): ZX-101A administered orally at level B once daily in a 28-day cycle
  Interventions: Drug: ZX-101A
- ZX-101A Dose Level C (Experimental): ZX-101A administered orally at level C once daily in a 28-day cycle
  Interventions: Drug: ZX-101A
- ZX-101A Dose Level D (Experimental): ZX-101A administered orally at level D once daily in a 28-day cycle
  Interventions: Drug: ZX-101A
- ZX-101A Dose Level E (Experimental): ZX-101A administered orally at level E once daily in a 28-day cycle
  Interventions: Drug: ZX-101A

INTERVENTIONS:
Drug: ZX-101A — Q.D., oral dosing

SUMMARY:
ZX-101A-201 is a phase I, open-label, multicenter study which includes dose escalation and dose expansion of ZX-101A. It is designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamic (PD), and antitumor activity of ZX-101A in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Phase I includes two parts: dose escalation and dose expansion.

* Part 1. ZX-101A dose escalation: 1) To evaluate the safety and tolerability of ZX-101A in patients with advanced solid tumors, and to determine the maximum tolerated dose (MTD) or optimal biological administration dose (OBD), and the recommended phase II dose clinical studies (RP2D); 2) To evaluate the pharmacokinetic (PK) characteristics of ZX-101A in patients with advanced solid tumors; 3) To evaluate the antitumor activity of ZX-101A in patients with advanced solid tumors, and provide dose basis for subsequent clinical trials; 4) To explore the pharmacodynamic (PD) characteristics of ZX-101A in patients with advanced solid tumors.
* Part 2. ZX-101A dose expansion: 1) To evaluate the safety and tolerability of ZX-101A in patients with advanced solid tumors; 2) To evaluate the PK profile of ZX-101A in patients with advanced solid tumors; 3) To evaluate the antitumor activity of ZX-101A in patients with advanced solid tumors, and provide dose basis for subsequent clinical trials; 4) To explore the PD characteristics of ZX-101A in patients with advanced solid tumors; 5) To explore the effect of ZX-101A on immune cytokines in serum.

ELIGIBILITY:
Inclusion Criteria:

* Males and females who are 18 to 75 years old.
* Minimum life expectancy ≥ 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Histologically or cytologically confirmed inoperable solid tumor subjects and failed standard treatment (PD during treatment or PD after last treatment), or subjects with advanced solid tumors or who cannot tolerate standard treatment and/or currently have no effective standard treatment.
* At least one measurable tumor lesion (according to RECIST V1.1 criteria).
* Systemic chemotherapy has been completed for at least 4 weeks (if the chemotherapy drugs are nitrosoureas and mitomycin C, it should be at least 6 weeks from the last chemotherapy); the anti-tumor monoclonal antibody treatment has been completed at least 4 weeks; small molecule targeted therapy has been completed at least 2 weeks or 5 half-lives of the drug (whichever is longer); Alternative treatment approved by the National Medical Products Administration (NMPA) has been completed for at least 4 weeks.
* Prior to the first dosing, radiotherapy has been completed for at least 4 weeks, local palliative radiotherapy has been completed for at least 2 weeks, and the acute toxicity caused by previous radiotherapy has recovered to ≤ grade 1.
* Prior cell or gene therapy was completed for at least 4 weeks before the first dose of study drug.
* Acceptable baseline assessment: 1) absolute neutrophil count (ANC) ≥1500 /mm3, platelet count (PLT)≥100K /mm3, and hemoglobin (Hb) ≥90 g/L for blood system (no blood transfusion and blood products or hematopoietic stimulating factor therapy within 14 day); 2) total bilirubin (TBIL) ≤1.5 × upper limit of normal (ULN) (≤3.0 × ULN in patients with Gilbert syndrome or liver metastases), alanine aminotransferase (ALT) ≤3.0×ULN, aspartate aminotransferase (AST) ≤3.0×ULN, and albumin ≥2.8 g/dL for liver function; 3) creatinine ≤1.5×ULN or creatinine clearance (Ccr) ≥50 ml/min (calculated according to Cockcroft-Gault formula, Ccr is calculated only when creatinine>1.5×ULN) for kidney function; 4) activated partial thromboplastin time (APTT) ≤1.5×ULN and international normalized ratio (INR) or prothrombin time (PT) ≤1.5×ULN for coagulation.
* Adverse reactions caused by previous treatment recovered to NCI-CTCAE V5.0 standard grade ≤1 before enrollment.
* Female subjects of childbearing age have negative serum pregnancy test results and agree to use effective contraception during the use of the study drug and within 6 months after the last dose.
* Men must agree to no sperm donations during the study and for 3 months after the last dose.
* Be able to understand the requirements of the study, willing to comply with all study procedures and sign the Institutional Review Board (IRB)-approved informed consent.

Exclusion Criteria:

* Previous use of PI3K δ/γ dual inhibitors.
* Received any anti-infective vaccine within 4 weeks before the first study drug.
* Received investigational study drug within 4 weeks or 5 half-lives, whichever is longer.
* History of other malignancy within the past 5 years, unless cured by surgery and sustained disease-free survival.
* Active autoimmune disease
* Have used systemic corticosteroids within 2 weeks before the first dosing.
* Serious medical conditions, including serious heart disease, uncontrolled diabetes, uncontrolled hypertension, active peptic ulcer, active bleeding, etc.
* Gastrointestinal dysfunction, including motility or malabsorption syndromes or inflammatory bowel disease which could limit absorption of study drug.
* Using medications that may lead to prolonged QT during the study period (e.g., antiarrhythmic drugs).
* Central nervous system or meningeal metastasis with clinical symptoms assessed by the investigator to be unsuitable for enrollment.
* Symptomatic ascites or pleural effusion or pericardial effusion.
* Current or past interstitial lung disease, hypersensitivity pneumonitis, pulmonary fibrosis, acute lung disease, etc.
* Active infection requiring systemic therapy.
* Active tuberculosis infection, receiving anti-tuberculosis treatment or received anti-tuberculosis treatment within 1 year before screening.
* Hepatitis B surface antigen (HBsAg) positive and HBV-DNA quantification > detection unit upper limit of normal value (ULN), hepatitis C antibody (HCV-Ab) positive and HCV-RNA quantification > detection unit upper limit of normal value, anti-human immunodeficiency virus antibody (Anti - HIV) positive, cytomegalovirus (CMV) infection or viremia, and active syphilis (any of the above). Hepatitis B virus subjects who are stable after 2 weeks of treatment (HBV-DNA quantification less than the lower limit of normal) and cured hepatitis C subjects (with known HCV history and with negative HCV RNA polymerase chain reaction [PCR] test results < 6 months prior to the start of ZX-101A administration) can be enrolled. CMV testing is required to confirm no CMV infection before screening.
* History of immunodeficiency, including a positive HIV test, or other acquired or congenital immunodeficiency disease, or a history of organ transplantation, or a history of allogeneic bone marrow transplantation, or a history of autologous hematopoietic stem cell transplantation.
* Received a major surgery or have not fully recovered from previous surgery within 4 weeks prior to the first dose of study drug.
* Uncontrolled or symptomatic hypercalcemia (>1.5 mmol/L ionized calcium or calcium >12 mg/dL or corrected serum calcium >ULN).
* In the judgment of the investigator, subjects are not suitable to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-03-09 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Defining the RP2D of ZX-101A | From Day 1 of Cycle 1 until 28 days after the last dose (up to 2 years). Each cycle is 28 days.
  To assess number of patients experiencing dose-limiting toxicities (DLTs)
To examine the incidence of clinical and laboratory adverse events after multiple doses of ZX-101A | From Day 1 of Cycle 1 until 28 days after the last dose (up to 2 years). Each cycle is 28 days.
  Incidence of treatment-emergent adverse events [safety and tolerability]

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  To evaluate the objective response rate (ORR) as determined by the specific disease response criteria
Duration of response (DoR) | Up to 2 years
  To examine the duration of response (DoR), defined as time from the date of first documentation of response to the date of the first documentation of progressive disease (PD), or death due to any cause
Progression free survival (PFS) | Up to 2 years
  To examine the the progression free survival (PFS), defined as time from the date of first dose of study treatment to the first date of documentation of PD, or death due to any cause
Disease control rate (DCR) | Up to 2 years
  To examine the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease to a therapeutic intervention
Overall survival (OS) | Up to 2 years
  To examine the overall survival (OS), defined as time from the date of first dose of study treatment to death due to any cause
Plasma Concentration of ZX-101A | Cycle1Day1 pre-dose and post-dose 0.5, 1, 2, 4, 6, 8, 24, 48, 72, 96 hours; Day18 and Day19 pre-dose; Day20 pre-dose and post-dose 0.5, 1, 2, 4, 6, 8 and 24hours; Cycle2Day1 pre-dose. Each cycle is 28 days.
  To assess the pharmacokinetic (PK) characteristics of ZX-101A in part 1
Plasma Concentration of ZX-101A | Cycle1Day13 and Day14 pre-dose; Day15 pre-dose and post-dose 0.5, 1, 2, 4, 6, 8, 24 hours; Cycle2Day1 pre-dose. Each cycle is 28 days.
  To assess the pharmacokinetic (PK) characteristics of ZX-101A in part 2
MDSC and CD8+ T cell levels in whole blood | Cycle1Day1, Cycle2Day1, Cycle3Day1. Each cycle is 28 days.
  To explore the pharmacodynamic (PD) characteristics of ZX-101A
Cytokines/chemokines levels in serum | Cycle1Day1, Cycle2Day1, Cycle3Day1. Each cycle is 28 days.
  To explore the pharmacodynamic (PD) characteristics of ZX-101A in part 2

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolin Qin, Ph.D, Study Director — Zenshine Pharmaceutical, Inc.
Locations (1):
- Beijing Cancer Hospital, Beijing, China